CLINICAL TRIAL: NCT02474446
Title: Determining the Effects of Race, Skin Colour and Genotype on the Response to Vitamin D Therapy
Brief Title: Getting Vitamin D Dosing Right
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH/14/053
Record Dates: First submitted 2015-06-04; First posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Vitamin D Status
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Anthropometry measurement, Skin colour grading using Fitzpatrick scale, Dietary intake of calcium and vitamin D using food frequency questionnaire (FFQ), Baseline fasting blood samples for vitamin D, VDBP, VDBP genotype, Calcium, Phosphorus, Albumin, Parathyroid Hormone(PTH), Alkaline Phosphatase, Bone turnover markers(P1NP, CTX).
  Fasting urine for Calcium Creatinine ratio. Saliva for bio-available Free Vitamin D measurement.
  Vitamin D administration under direct supervision. Spot Urine sample for calcium : creatinine ratio after a week. Repeat all measurements done at baseline except VDBP genotype 4 weeks from baseline.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 150,000 IU of Vitamin D3 Oral solution

SUMMARY:
The investigators want to make sure that people get the right dose of Vitamin D treatment. They will therefore investigate how skin colour, body mass index, ethnicity, vitamin D binding protein and genetic variation affect the response to a standard course of vitamin D in young adults, as a prelude to further studies in younger children.

DETAILED DESCRIPTION:
The Department of Health and the Chief Medical Officer have identified vitamin D deficiency as a key area of interest and concern for public health.

The main function of vitamin D is to enable dietary calcium to be absorbed from the intestine. Low levels of vitamin D can lead to diseases of bone such as rickets and osteomalacia and are linked to a higher risk of fracturing bones in older women with osteoporosis.

Vitamin D levels may be affected by the skin colour, body mass index (BMI), lifestyle or environment in which someone lives, and by their genetic makeup. Vitamin D levels tend to be lower in people with higher BMI and / or darker coloured skin or if the skin is covered by clothing because a lot of vitamin D is made from the action of sunlight on natural chemicals in the skin.

Vitamin D does occur naturally in the diet in foods like oily fish, and also vitamin D can be given as a supplement either on its own or as part of a multivitamin tablet.

There is natural variation from one person to another in how well the system controlling vitamin D blood levels works. Vitamin D circulates bound to a carrier protein, vitamin D binding protein (VDBP). When vitamin D levels are measured, both vitamin D bound to the protein and "free" vitamin D are measured.

A recent study in America showed that when "free" vitamin D levels (total vitamin D minus vitamin D bound to VDBP) are measured, they correlate very closely with other factors that help determine blood calcium levels.This variation is determined in part by a person's genetic makeup, and recent large studies have identified specific genetic variations that are linked to blood levels of vitamin D; some of these vary with the person's ethnic origin.

At present if someone has low vitamin D levels that put them at increased risk of bone problems, a course of vitamin D treatment is given.

When the investigators assessed their regular treatment given to children recently, they found some individuals developed very high blood vitamin D levels and others didn't.

They don't know how VDBP levels affect the response to treatment with vitamin D.

Further variation can occur because of the distribution of vitamin D into fat tissue. The investigators will measure height and weight, and waist and hip circumference and calculate Body Mass Index, body surface area (BSA) and waist: hip ratio as proxy measures of fat mass.

They will also evaluate whether blood or saliva tests give better information about vitamin D levels. The information about how these factors affect the response to vitamin D will help the clinicians choose the right dose of vitamin D for studies in younger children who are still growing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young male adults aged 18 25 years
* Free from any condition affecting bone health, general nutrition, growth and glucose metabolism.

Exclusion Criteria:

* Subjects with any chronic illness involving the liver and kidney
* Use of steroids, anticonvulsants or any medication that might affect calcium and vitamin D metabolism.
* Potential participants who have made plans to travel abroad during the study period.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Increase in serum 25 hydroxyvitaminD (25OHD) levels | Participants will be followed for the duration of the study, an expected average of 4 weeks
  Increase in serum 25OHD levels by at least 25 nmol/L in the majority of the participants, 4 weeks after administration of 150,000 units of vitamin D, according to genotype and ethnicity.

SECONDARY OUTCOMES:
Determine if dark skin colour or South Asian heritage reduces the increase in serum 25OHD. | Participants will be followed for the duration of the study, an expected average of 4 weeks
  Change in serum 25OHD 4 weeks after dosing with 150,000 international units(IU) of Vitamin D according to skin colour
  Change in urinary calcium:creatinine ratio at 1 week after dosing. Change in in serum calculated free vitamin D, calcium, PTH and alkaline phosphatase 4 weeks after dosing.
Change in serum calculated free vitamin D | Participants will be followed for the duration of the study, an expected average of 4 weeks
  Change in calculated 'free' 25OHD 4 weeks after dosing with 150,000IU of Vitamin D
  Change in urinary calcium:creatinine ratio at 1 week after dosing. Change in in serum calculated free vitamin D, calcium, PTH and alkaline phosphatase 4 weeks after dosing.
Determine if variation in Group specific component(GC) genotype is associated with variation in the increase in serum 25OHD. | Participants will be followed for the duration of the study, an expected average of 4 weeks
  Change in serum 25OHD levels according to GC Genotype
Determine the extent of parathyroid hormone (PTH) suppression in relation to overall increases in total and free serum 25OHD | Participants will be followed for the duration of the study, an expected average of 4 weeks
  Extent of PTH suppression before and after dosing with 150,000IU of Vitamin D

OTHER OUTCOMES:
Evidence of hypercalciuria | Participants will be followed for the duration of the study, an expected average of 4 weeks
  Spot urine calcium:creatinine ratio will be performed on second void fasting urine 1 week after dosing to reassure that no hypercalciuria has occurred in any subject.

CONTACTS AND LOCATIONS:
Overall Officials: Sujatha Gopal, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom